CLINICAL TRIAL: NCT02946996
Title: Randomized Phase II Study of Pharmacologic Manipulation of AGE (Advanced Glycation Endproducts) Levels in Prostate Cancer Patients Receiving Androgen Deprivation Therapy
Brief Title: Study of Pharmacologic Manipulation of AGE (Advanced Glycation Endproducts) Levels in Prostate Cancer Patients Receiving Androgen Deprivation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator retired from clinical practice prior to enrollment goal being met.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102508
Record Dates: First submitted 2016-10-18; First posted 2016-10-27 (Estimated); Results first posted 2025-02-03 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Metformin Only (Experimental): Subjects will be supplied with metformin tablets850mg. During the ramp up phase subjects will take metformin in the morning. During weeks 2-12 the metformin tablet will be taken approximately 12 hours apart.
  Interventions: Drug: Metformin
- OPC Only (Experimental): Subjects will take one OPC capsule at the same time each morning and evening, approximately 12 hours apart during weeks 1-12.
  Interventions: Other: OPC
- Metformin plus OPC (Experimental): During week 1, subjects will take one metformin tablet in the morning and one OPC tablet in the morning and in the evening, about12 hours apart.
  During weeks 2-12 the metformin tablet will betaken approximately 12 hours apart and one OPC about 12 hours apart, in the morning and in the evening.
  Interventions: Drug: Metformin; Other: OPC

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin Only; Metformin plus OPC
Other: OPC — OPC is a derivative of grape seed extract
  Arms: Metformin plus OPC; OPC Only

SUMMARY:
The purpose of this study is to look at the effect that the study drug OPC has on AGE levels in patients with prostate cancer.

DETAILED DESCRIPTION:
AGEs are a type of metabolite, or substance, found in the food. The AGE content in food is determined by the types of food you eat and also how you prepare your food. The researchers helping conduct this study have found a potential link between AGE levels and cancer. The purpose of this study is to see if Oligomeric Procyanidin Complex (OPC) has an effect on the AGE levels in your blood and to see if those AGE levels have an effect on your cancer.

ELIGIBILITY:
Inclusion Criteria

1. Confirmation of adenocarcinoma of the prostate that is documented by one of the following: pathology report or clinic note with documented history of prostate cancer.
2. Subjects must be receiving ADT with a GnRH agonist or antagonist, with or without an anti-androgen, with a current testosterone level documented to be <50ng/dL at enrollment. Subjects whose ADT is interrupted may enroll or continue on study as long as the testosterone is documented to remain <50ng/dL for the entire duration of study participation. Subjects who have undergone orchiectomy are also eligible.
3. Prior cytotoxic chemotherapy for metastatic prostate cancer; prior treatment with genomically-targeted agents, or Provenge is allowed.
4. Subjects must have adequate hematologic, renal, and hepatic function at baseline, as follows:

   * Hematology parameters: ANC >1000/mcL, platelets > 100,000/mcL, Hgb >8.0gm/dL
   * Renal Function: eGFR of > 45mls/min using Cockgroft and Gault formula (see appendix C).
   * Liver Function: Total bilirubin ≤ULN, AST and ALT <1.5xULN
5. Able to swallow and retain oral medication
6. ECOG performance status of 0 - 2
7. Ability to sign written informed consent
8. Testosterone level <50ng/dL

Exclusion Criteria

1. Known allergy to grapes or grape seed
2. History of receiving more than 2 classes of ADT.
3. Current use of strong antioxidants (extracts from grape seed, milk thistle; pine bark, green tea, saw palmetto; resveratrol; flavonoids; catechins; ellagic acid), large quantities of red grapes, white button mushrooms, red wine. See section 4.7 for more details.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 14 non-evaluable
Groups:
- Metformin Only: Subjects will be supplied with metformin tablets850mg. During the ramp up phase subjects will take metformin in the morning. During weeks 2-12 the metformin tablet will be taken approximately 12 hours apart.
  Metformin
- Metformin Plus OPC: During week 1, subjects will take one metformin tablet in the morning and one OPC tablet in the morning and in the evening, about12 hours apart.
  During weeks 2-12 the metformin tablet will betaken approximately 12 hours apart and one OPC about 12 hours apart, in the morning and in the evening.
  Metformin
  OPC: OPC is a derivative of grape seed extract
Period: Overall Study
Arm/Group | Metformin Only | OPC Only | Metformin Plus OPC
Started | 12 | 16 | 13
Completed | 9 | 10 | 8
Not Completed | 3 | 6 | 5
Not completed — non-evaluable | 3 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Only | OPC Only | Metformin Plus OPC | Total
Number analyzed (Participants) | 12 | 16 | 13 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (6.1) | 73.6 (5.0) | 74.9 (7.8) | 73.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 12 | 16 | 13 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/AA | 5 | 1 | 2 | 8
  White | 7 | 15 | 11 | 33
Region of Enrollment [Number; unit: participants]
  United States | 12 | 16 | 13 | 41

OUTCOME MEASURES:

1. Primary Outcome: AGE Level Reduction
Description: The primary objective is to determine if any of the test agent are able to reduce AGE levels by an average of 30% (or greater) in 50% or more of test subjects.
Time Frame: 85 days
Measure: Median (30% Confidence Interval); unit: ng/ml
Arm/Group | Metformin Only | OPC Only | Metformin Plus OPC
Number analyzed (Participants) | 8 | 10 | 9
ng/ml | 1.49 [-1.51 to 4.52] | 0.49 [-3.32 to 1.18] | 0.8 [-0.88 to 3.09]

2. Secondary Outcome: Correlation Between Changes to AGE Level and Changes to PSA
Time Frame: 85 days
Reporting Status: Not Posted

3. Secondary Outcome: Correlation Between Changes to AGE Level and Changes to BMI
Time Frame: 85 days
Reporting Status: Not Posted

4. Secondary Outcome: Correlation Between Changes to AGE Level and Changes to Insulin Resistance (HOMA-IR)
Time Frame: 85 days
Reporting Status: Not Posted

5. Secondary Outcome: Correlation Between Changes to AGE Level and Changes to A1C.
Time Frame: 85 days
Reporting Status: Not Posted

6. Secondary Outcome: Correlations Between Changes to AGE Level and Changes to Testosterone.
Time Frame: 85 days
Reporting Status: Not Posted

7. Secondary Outcome: Correlation Between Changes to AGE Level and Changes to Lipids.
Time Frame: 85 days
Reporting Status: Not Posted

8. Secondary Outcome: Correlation Between Changes to AGE Level and Changes to Diet.
Time Frame: 85 days
Reporting Status: Not Posted

9. Secondary Outcome: Correlation Between Changes to AGE Level and Changes to Quality of Life
Time Frame: 85 days
Reporting Status: Not Posted

10. Secondary Outcome: Frequency of Adverse Events as Assessed by CTCAE v. 4
Description: Toxicities will be tabulated per arm by type and grade and the proportion of patients with grade 3, grade 4 or an SAE will be estimated with a 90% confidence interval.
Time Frame: 85 days
Reporting Status: Not Posted

11. Secondary Outcome: Correlation Between AGE Levels and Plasma IL6
Time Frame: 85 days
Reporting Status: Not Posted

12. Secondary Outcome: Correlation Between AGE Levels and Leptin
Time Frame: 85 days
Reporting Status: Not Posted

13. Secondary Outcome: Correlation Between AGE Levels and C-reactive Protein (CRP)
Time Frame: 85 days
Reporting Status: Not Posted

14. Secondary Outcome: Correlation Between AGE Levels and Malondialdehyde (MDA)
Time Frame: 85 days
Reporting Status: Not Posted

15. Secondary Outcome: Correlation Between AGE Levels and oxLDLs (Low Density Lipoprotein)
Time Frame: 85 days
Reporting Status: Not Posted

16. Secondary Outcome: Correlation Between AGE Levels and sRAGE (Soluble Receptor for AGE)
Time Frame: 85 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 85 Days
Arm/Group | Metformin Only | OPC Only | Metformin Plus OPC
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 9/12 | 4/16 | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin Only (N=12) | OPC Only (N=16) | Metformin Plus OPC (N=13)
abdominal pain (Gastrointestinal disorders) | 7 (16) | 1 (1) | 7 (17) — nausea, diarrhea, bloating
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) — Headache
broken tooth (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
weight loss (Investigations) | 1 (1) | 0 (0) | 2 (2)
flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2)
Libido Decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hot Flashes (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) — Pruritis, hyperhydrosis
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) — Upper respiratory infection
knee swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
R ankle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) — gout
non cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT02946996/Prot_SAP_000.pdf